CLINICAL TRIAL: NCT01354431
Title: A Randomized, Blinded, Phase 2 Dose-Ranging Study Of BMS-936558 (MDX-1106) In Subjects With Progressive, Advanced/Metastatic Clear-Cell Renal Cell Carcinoma Who Have Received Prior Anti-Angiogenic Therapy
Brief Title: BMS-936558 (MDX-1106) In Subjects With Advanced/Metastatic Clear-Cell Renal Cell Carcinoma (RCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharma USA Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CA209-010
Expanded Access: NCT03126643 (Approved for marketing)
Record Dates: First submitted 2011-05-10; First posted 2011-05-16 (Estimated); Results first posted 2015-10-20 (Estimated); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Renal Cell Carcinoma
Keywords: Advanced/Metastatic; clear cell component
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — Nivolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: nivolumab - 0.3 mg/kg (Experimental)
  Interventions: Biological: nivolumab
- Arm 2: nivolumab - 2.0 mg/kg (Experimental)
  Interventions: Biological: nivolumab
- Arm 3: nivolumab - 10.0 mg/kg (Experimental)
  Interventions: Biological: nivolumab

INTERVENTIONS:
Biological: nivolumab — Solution, Intravenous (IV), 0.3 mg/kg, every 3 weeks (Q 3 weeks), Until Progressive disease (PD), toxicity or discontinue for other reasons
  Other Names: BMS-936558
  Arms: Arm 1: nivolumab - 0.3 mg/kg
Biological: nivolumab — Solution, Intravenous (IV), 2.0 mg/kg, every 3 weeks (Q 3 weeks), Until Progressive disease (PD), toxicity or discontinue for other reasons
  Other Names: BMS-936558
  Arms: Arm 2: nivolumab - 2.0 mg/kg
Biological: nivolumab — Solution, Intravenous (IV), 10.0 mg/kg, every 3 weeks (Q 3 weeks), Until Progressive disease (PD), toxicity or discontinue for other reasons
  Other Names: BMS-936558
  Arms: Arm 3: nivolumab - 10.0 mg/kg

SUMMARY:
The purpose of this study is to measure how active BMS-936558 (nivolumab) is against Renal Cell Carcinoma (RCC) as measured by the disease not progressing and whether a dose response relationship exists.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of Renal cell carcinoma (RCC) with a clear cell component
* Previous treatment with at least one anti-angiogenic agent
* Progressed within 6 months of study enrollment
* Subjects should not have had more than 3 prior treatments for locally advanced or metastatic disease
* Must have available tumor tissue for submission
* Subjects must also meet various laboratory parameters for inclusion

Exclusion Criteria:

* Subjects with any active autoimmune disease or a history of known autoimmune disease

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2011-05-31 (Actual); Primary Completion 2013-05-15 (Actual); Study Completion 2021-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (41):
- United States (34):
  - UCSD Moores Cancer Center, La Jolla, California
  - Ucla, Los Angeles, California
  - Samuel Oschin Comprehensive Cancer Inst., Los Angeles, California
  - Stanford Cancer Center, Stanford, California
  - University Of Colorado, Aurora, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Northwestern University Feinberg School Of Medicine, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana University Health Melvin And Bren Simon Cancer Center, Indianapolis, Indiana
  - University Of Kansas Medical Center, Kansas City, Kansas
  - University Of Maryland, Baltimore, Maryland
  - The Bunting-Blaustein Cancer Research Building, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Ctr., Boston, Massachusetts
  - University Of Michigan Medical Center, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Masonic Cancer Ctr, University Of Minnesota, Minneapolis, Minnesota
  - North Mississippi Hematology And Oncology Associates, Ltd, Tupelo, Mississippi
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - St. Luke'S Roosevelt Hospital Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Memorial Sloan Kettering Nassau, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Blumenthal Cancer Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University Of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University Of South Carolina, Charleston, South Carolina
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Ctr, Nashville, Tennessee
  - University of Washington - Seattle Cancer Care Alliance, Seattle, Washington
  - Wheaton Franciscan Health Care, Wauwatosa, Wisconsin
- Canada (5):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Centre D'Oncologie Dr-Leon-Richard, Moncton, New Brunswick
  - Local Institution, Halifax, Nova Scotia
  - London Regional Cancer Program, London, Ontario
  - Centre Hospitalier Universitaire De Montreal-Notre-Dame Hosp, Montreal, Quebec
- Local Institution, Helsinki, Finland
- Local Institution, Siena, Italy

REFERENCES:
- [Derived] George S, Motzer RJ, Hammers HJ, Redman BG, Kuzel TM, Tykodi SS, Plimack ER, Jiang J, Waxman IM, Rini BI. Safety and Efficacy of Nivolumab in Patients With Metastatic Renal Cell Carcinoma Treated Beyond Progression: A Subgroup Analysis of a Randomized Clinical Trial. JAMA Oncol. 2016 Sep 1;2(9):1179-86. doi: 10.1001/jamaoncol.2016.0775. PMID 27243803
- [Derived] Motzer RJ, Rini BI, McDermott DF, Redman BG, Kuzel TM, Harrison MR, Vaishampayan UN, Drabkin HA, George S, Logan TF, Margolin KA, Plimack ER, Lambert AM, Waxman IM, Hammers HJ. Nivolumab for Metastatic Renal Cell Carcinoma: Results of a Randomized Phase II Trial. J Clin Oncol. 2015 May 1;33(13):1430-7. doi: 10.1200/JCO.2014.59.0703. Epub 2014 Dec 1. PMID 25452452
- [Derived] George S, Pili R, Carducci MA, Kim JJ. Role of immunotherapy for renal cell cancer in 2011. J Natl Compr Canc Netw. 2011 Sep 1;9(9):1011-8. doi: 10.6004/jnccn.2011.0085. PMID 21917625
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 168 participants were randomized, 167 participants were treated.
Groups:
- Nivolumab 0.3 mg/kg: Nivolumab 0.3 mg/kg IV Q3W
- Nivolumab 2 mg/kg: Nivolumab 2 mg/kg IV Q3W
- Nivolumab 10 mg/kg: Nivolumab 10 mg/kg IV Q3W
Period: Pre-Treatment Period
Arm/Group | Nivolumab 0.3 mg/kg | Nivolumab 2 mg/kg | Nivolumab 10 mg/kg
Started | 60 | 54 | 54
Completed (Completed = Moved to Treatment Period) | 59 | 54 | 54
Not Completed | 1 | 0 | 0
Not completed — Not reported | 1 | 0 | 0
Period: Treatment Period
Arm/Group | Nivolumab 0.3 mg/kg | Nivolumab 2 mg/kg | Nivolumab 10 mg/kg
Started | 59 | 54 | 54
Completed | 0 | 0 | 0
Not Completed | 59 | 54 | 54
Not completed — Disease Progression | 50 | 40 | 44
Not completed — Study Drug Toxicity | 5 | 8 | 4
Not completed — Death | 0 | 1 | 0
Not completed — AE unrelated to study drug | 1 | 2 | 5
Not completed — Participant request to discontinue | 2 | 2 | 1
Not completed — Participant withdrew consent | 0 | 1 | 0
Not completed — Participant no longer meeting study criteria | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Randomized participants were included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab 0.3 mg/kg | Nivolumab 2 mg/kg | Nivolumab 10 mg/kg | Total
Number analyzed (Participants) | 60 | 54 | 54 | 168
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 37 | 41 | 35 | 113
  >=65 years | 23 | 13 | 19 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (8.8) | 60.8 (8.2) | 60.6 (9.6) | 60.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 14 | 14 | 47
  Male | 41 | 40 | 40 | 121
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 53 | 53 | 54 | 160
  Unknown or Not Reported | 7 | 1 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from randomization to date of first disease progression (either clinical or radiographic progression, as assessed by the investigator). Tumor assessments (radiographic scans) were done every 6 weeks from randomization for the first 12 months, then every 12 weeks until progression. Survival was assessed every 3 months. The analysis of PFS was conducted after approximately 116 events (progression or death), approximately 2 years. PFS was calculated based on investigator's assessment of first date of progression (either clinical or radiographic progression) or date of death if progression did not occur. Progression was at least a 20% increase in the sum of diameters of the longest target lesions since screening (the sum must be an absolute increase of at least 5 mm), or measurable increase in non-target lesion or appearance of one or more new lesions.
Time Frame: From randomization to disease progression or death (up to approximately 2 years)
Population: All randomized participants
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Nivolumab 0.3 mg/kg | Nivolumab 2 mg/kg | Nivolumab 10 mg/kg
Number analyzed (Participants) | 60 | 54 | 54
Months | 2.63 [1.81 to 3.02] | 4.11 [2.86 to 5.39] | 4.17 [2.79 to 5.49]

2. Secondary Outcome: Best Overall Response Rate (BORR)
Description: BORR is defined as the percentage of participants whose best response is either partial response (PR) or complete response (CR). Tumor response was evaluated by investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
  CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  PR: at least 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  80% confidence interval is based on the Clopper and Pearson method
Time Frame: From randomization until disease progression or discontinuation of study therapy (up to approximately 2 years)
Population: All randomized participants
Measure: Number (80% Confidence Interval); unit: Percent of participants
Arm/Group | Nivolumab 0.3 mg/kg | Nivolumab 2 mg/kg | Nivolumab 10 mg/kg
Number analyzed (Participants) | 60 | 54 | 54
Percent of participants | 20.0 [13.4 to 28.2] | 24.1 [16.6 to 33.1] | 20.4 [13.4 to 29.1]

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from date of randomization until date of death. If the participant did not die, overall survival will be censored on the last date the participant was known to be alive. Survival status is collected at each visit during treatment and every 3 months during follow-up.
  OS is based on Kaplan-Meier estimates.
Time Frame: From randomization to to date of death (up to approximately 8 years)
Population: All randomized participants
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Nivolumab 0.3 mg/kg | Nivolumab 2 mg/kg | Nivolumab 10 mg/kg
Number analyzed (Participants) | 60 | 54 | 54
Months | 18.45 [16.23 to 23.98] | 25.46 [19.78 to 31.24] | 24.82 [15.31 to 25.95]

4. Secondary Outcome: Number of Participants Experiencing Adverse Events
Description: Number of participants experiencing different types of events, including Adverse Events (AEs), Drug-related AEs, AEs leading to discontinuation, Drug-related AEs leading to discontinuation, Serious Adverse Events (SAEs), Drug-related SAEs.
  Events are classified based on the NCI Common Terminology Criteria (CTC) version 4.0
Time Frame: From first dose to 30 days following last dose (up to approximately 6 years)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab 0.3 mg/kg | Nivolumab 2 mg/kg | Nivolumab 10 mg/kg
Number analyzed (Participants) | 59 | 54 | 54
Participants
  Any AEs | 58 | 54 | 53
  Drug-related AEs | 44 | 36 | 41
  AEs leading to discontinuation | 6 | 10 | 10
  Drug-related AEs leading to discontinuation | 4 | 5 | 4
  SAEs | 26 | 26 | 22
  Drug-related SAEs | 3 | 4 | 3

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from first dose to study completion date (up to approximately 118 months). SAEs and NSAEs were assessed from first dose to 100 days following last dose (up to approximately 79 months).
Description: All-cause mortality: all randomized participants SAEs and NSAEs: all treated participants
Arm/Group | NIVOLUMAB 0.3 mg/kg | NIVOLUMAB 2 mg/kg | NIVOLUMAB 10 mg/kg
All-Cause Mortality (participants affected / at risk) | 51/60 | 46/54 | 47/54
Serious Adverse Events (participants affected / at risk) | 30/59 | 35/54 | 24/54
Other Adverse Events (participants affected / at risk) | 55/59 | 54/54 | 52/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NIVOLUMAB 0.3 mg/kg (N=59) | NIVOLUMAB 2 mg/kg (N=54) | NIVOLUMAB 10 mg/kg (N=54)
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0
Goitre (Endocrine disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Small intestine ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Death (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0
Localised oedema (General disorders) | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 2 | 1
Pain (General disorders) | 2 | 0 | 1
Pyrexia (General disorders) | 0 | 2 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Gallbladder obstruction (Hepatobiliary disorders) | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Biliary sepsis (Infections and infestations) | 1 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Cholecystitis infective (Infections and infestations) | 0 | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 3 | 2
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Influenza B virus test positive (Investigations) | 1 | 0 | 0
Liver function test increased (Investigations) | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 2
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 5 | 3
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 1
Central nervous system lesion (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0
Hemianopia homonymous (Nervous system disorders) | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 2 | 0
Paralysis recurrent laryngeal nerve (Nervous system disorders) | 1 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 2 | 1 | 0
Spinal cord compression (Nervous system disorders) | 2 | 4 | 0
Device failure (Product Issues) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Urogenital haemorrhage (Renal and urinary disorders) | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Knee arthroplasty (Surgical and medical procedures) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NIVOLUMAB 0.3 mg/kg (N=59) | NIVOLUMAB 2 mg/kg (N=54) | NIVOLUMAB 10 mg/kg (N=54)
Anaemia (Blood and lymphatic system disorders) | 9 | 8 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3 | 0
Palpitations (Cardiac disorders) | 3 | 0 | 1
Tachycardia (Cardiac disorders) | 3 | 1 | 3
Deafness (Ear and labyrinth disorders) | 0 | 1 | 3
Hypothyroidism (Endocrine disorders) | 3 | 3 | 5
Vision blurred (Eye disorders) | 0 | 0 | 3
Abdominal distension (Gastrointestinal disorders) | 3 | 3 | 2
Abdominal pain (Gastrointestinal disorders) | 5 | 4 | 5
Abdominal pain upper (Gastrointestinal disorders) | 2 | 4 | 4
Constipation (Gastrointestinal disorders) | 13 | 19 | 11
Diarrhoea (Gastrointestinal disorders) | 9 | 10 | 16
Dry mouth (Gastrointestinal disorders) | 4 | 3 | 7
Dyspepsia (Gastrointestinal disorders) | 3 | 3 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 3 | 3
Flatulence (Gastrointestinal disorders) | 1 | 0 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 4
Nausea (Gastrointestinal disorders) | 16 | 15 | 12
Stomatitis (Gastrointestinal disorders) | 3 | 4 | 0
Toothache (Gastrointestinal disorders) | 2 | 1 | 3
Vomiting (Gastrointestinal disorders) | 12 | 8 | 10
Asthenia (General disorders) | 1 | 3 | 3
Chest discomfort (General disorders) | 1 | 0 | 4
Chest pain (General disorders) | 1 | 3 | 1
Chills (General disorders) | 4 | 5 | 7
Fatigue (General disorders) | 25 | 25 | 29
Influenza like illness (General disorders) | 1 | 2 | 4
Mucosal inflammation (General disorders) | 2 | 0 | 3
Oedema (General disorders) | 3 | 3 | 1
Oedema peripheral (General disorders) | 14 | 10 | 11
Pain (General disorders) | 3 | 4 | 2
Pyrexia (General disorders) | 6 | 9 | 6
Hypersensitivity (Immune system disorders) | 2 | 1 | 9
Bronchitis (Infections and infestations) | 3 | 1 | 3
Nasopharyngitis (Infections and infestations) | 1 | 1 | 3
Rhinitis (Infections and infestations) | 3 | 1 | 1
Sinusitis (Infections and infestations) | 7 | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 7 | 11 | 8
Urinary tract infection (Infections and infestations) | 2 | 4 | 2
Contusion (Injury, poisoning and procedural complications) | 3 | 1 | 3
Fall (Injury, poisoning and procedural complications) | 3 | 3 | 2
Alanine aminotransferase increased (Investigations) | 4 | 4 | 3
Aspartate aminotransferase increased (Investigations) | 4 | 5 | 3
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 5
Blood creatinine increased (Investigations) | 7 | 3 | 2
Weight decreased (Investigations) | 9 | 7 | 9
Weight increased (Investigations) | 7 | 3 | 5
Decreased appetite (Metabolism and nutrition disorders) | 8 | 15 | 11
Dehydration (Metabolism and nutrition disorders) | 3 | 6 | 6
Hypercalcaemia (Metabolism and nutrition disorders) | 4 | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 7 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 5 | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 18 | 16
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 17 | 17
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 2 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 8 | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 5 | 9
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 16 | 5
Dizziness (Nervous system disorders) | 8 | 5 | 7
Dysarthria (Nervous system disorders) | 0 | 0 | 3
Headache (Nervous system disorders) | 7 | 6 | 9
Hypoaesthesia (Nervous system disorders) | 1 | 4 | 1
Neuropathy peripheral (Nervous system disorders) | 2 | 2 | 5
Paraesthesia (Nervous system disorders) | 2 | 2 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 2 | 5
Taste disorder (Nervous system disorders) | 1 | 0 | 4
Anxiety (Psychiatric disorders) | 3 | 4 | 4
Depression (Psychiatric disorders) | 2 | 2 | 5
Insomnia (Psychiatric disorders) | 6 | 8 | 3
Haematuria (Renal and urinary disorders) | 2 | 1 | 3
Pollakiuria (Renal and urinary disorders) | 3 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 20 | 11
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 11 | 10
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 3
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 6 | 10
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 4 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 4 | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 7 | 9
Rash (Skin and subcutaneous tissue disorders) | 8 | 6 | 12
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 5 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 3
Flushing (Vascular disorders) | 0 | 4 | 3
Hot flush (Vascular disorders) | 0 | 3 | 3
Hypertension (Vascular disorders) | 3 | 3 | 4
Hypotension (Vascular disorders) | 0 | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.